CLINICAL TRIAL: NCT05879614
Title: An Open-Label Study of the Safety, Tolerability, and Pharmacokinetics of Oral NNZ-2591 in Prader-Willi Syndrome (PWS-001)
Brief Title: An Open-Label Study of Oral NNZ-2591 in Prader-Willi Syndrome (PWS-001)
Acronym: PWS-001
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Revised development strategy
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-2591-PWS-001
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — cyclo-L-glycyl-L-2-allylproline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNZ-2591 (Experimental): NNZ-2591 oral solution (50mg/mL) to be administered twice daily for 13 weeks.
  Interventions: Drug: NNZ-2591

INTERVENTIONS:
Drug: NNZ-2591 — NNZ-2591 oral solution (50mg/mL) to be administered twice daily for 13 weeks.
  Other Names: Cyclo-L-Glycyl-L-2-Allylproline

SUMMARY:
A study of the safety, tolerability and pharmacokinetics of NNZ-2591 and measures of efficacy in children and adolescents with Prader-Willi Syndrome.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate the safety, tolerability and pharmacokinetics of treatment with NNZ-2591 oral solution in children and adolescents with Prader-Willi Syndrome. The secondary purpose is to investigate measures of efficacy. Subjects will receive treatment with NNZ-2591 oral solution (50 mg/mL) doses for a total of 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PWS with a documented disease-causing genetic abnormality of the chromosome 15q11-q13 confirmed by DNA methylation and microarray.
2. Males or females aged 4-12 years, inclusive.
3. Body weight of 12 kg to 100kg (inclusive) at Baseline.
4. Subjects with a Clinical Global Impression - Severity (CGI-S) score of 4 or greater at the Screening visit.
5. Must currently be on treatment with growth hormone.
6. Each subject must be able to swallow the study medication provided as a liquid solution.
7. Caregiver(s) must have sufficient English language skills.
8. Subject and caregiver must reside in the US and have been resident in the US for at least 3 months prior to screening.

Exclusion Criteria:

1. Body weight <12 kg or >100 kg at Baseline.
2. HbA1c values above 7% at the Screening visit.
3. Clinically significant abnormalities in safety laboratory tests and vital signs at Screening.
4. Positive pregnancy test at the Screening visit.
5. Positive drugs of abuse screen not explained by concomitant medications.
6. Abnormal QTcF interval or prolongation at Screening.
7. Any other clinically significant finding on ECG at the Screening visit.
8. Positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening or Baseline.
9. Previous COVID 19 infection with last 12 months that required hospitalization.
10. Previous COVD-19 infection involving multi-organ systems, resulting in Multisystem Inflammatory Syndrome in Children (MIS-C) or with clinically significant long term effects.
11. COVID-19 infection associated with acute kidney injury (AKI) or renal conditions.
12. Renal conditions or abnormalities identified in laboratory testing, imaging or medical history.
13. Liver conditions and Hepatic abnormalities.
14. Vision abnormalities and Ocular conditions.
15. Excluded concomitant treatments.
16. Unstable seizure profile.
17. Current clinically significant cardiovascular, gastrointestinal, or respiratory disease, or clinically significant organ impairment, or endocrine disease with the exception of obesity and controlled hypothyroidism.
18. Current clinically significant hypo or hyperthyroidism, Type 1 or Type 2 diabetes mellitus requiring insulin (whether well controlled or uncontrolled), or uncontrolled Type 1 or Type 2 diabetes.
19. Has planned surgery during the study.
20. History of, or current, cerebrovascular disease or brain trauma.
21. History of, or current catatonia or catatonia-like symptoms.
22. History of, or current, malignancy.
23. Current major or persistent depressive disorder (including bipolar depression).
24. Significant uncorrected hearing impairment.
25. Allergy to strawberry.
26. Has participated in another interventional clinical study within 30 days prior to start of Screening.
27. Subject is judged by the Investigator or Medical Monitor to be inappropriate for the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 13 weeks
  To examine the incidence, severity and frequency of adverse events (AEs), including serious adverse events (SAEs) during treatment with NNZ-2591.
Pharmacokinetic - Measurement of Cmax | 13 weeks
  Maximum observed concentration (Cmax) of NNZ-2591
Pharmacokinetic - Measurement of AUC | 13 weeks
  Area under the concentration-time curve of NNZ-2591
Pharmacokinetic - Measurement of time to Cmax | 13 weeks
  Time to Cmax of NNZ-2591
Pharmacokinetic - Measurement of t1/2 | 13 weeks
  Apparent terminal elimination half-life of NNZ-2591

SECONDARY OUTCOMES:
Exploratory efficacy measurement | 13 weeks
  Assessed by PWS-specific Clinical Global Impression Scale & Domain -Overall Improvement Score (CGI-I)
Exploratory efficacy measurement | 13 weeks
  Assessed by Caregiver Global Impression-Change Score
Exploratory efficacy measurement | 13 weeks
  Assessed by PWS-specific Clinical Global Impression Scale-Severity (CGI-S) Overall Score
Exploratory efficacy measurement | 13 weeks
  Assessed by Caregiver Top 3 Concerns Likert Scale Scores
Exploratory efficacy measurement | 13 weeks
  Assessed by PWS Profile Score
Exploratory efficacy measurement | 13 weeks
  Assessed by PWS Anxiousness and Distress Behaviors Questionnaire Score (PADQ)
Exploratory efficacy measurement | 13 weeks
  Assessed by Autism Diagnostic Observation Schedule (ADOS-2), Repetitive behaviors and Social scores
Exploratory efficacy measurement | 13 weeks
  Assessed by Hyperphagia Questionnaire-Clinical Trials (HQ-CT) Score
Exploratory efficacy measurement | 13 weeks
  Assessed by Food Safety Zone Questionnaire Score
Exploratory efficacy measurement | 13 weeks
  Assessed by Vineland Adaptive Behavior Scales-3 Growth Scale Scores
Exploratory efficacy measurement | 13 weeks
  Assessed by Zarit Burden Interview Score
Exploratory efficacy measurement | 13 weeks
  Assessed by Child Sleep Habits Questionnaire (CSHQ)
Exploratory efficacy measurement | 13 weeks
  Assessed by Impact of Childhood Neurological Disability Scale (ICND)
Exploratory efficacy measurement | 13 weeks
  Assessed by Quality of Life Inventory-Disability (QI-Disability)
Exploratory efficacy measurement | 13 weeks
  Assessed by Kaufman Brief Intelligence Test or Mullen Scales of Early Learning
Exploratory efficacy measurement | 13 weeks
  Assessed by PWS Suicidality Assessment
Exploratory efficacy measurement | 13 weeks
  Assessed by Caregiver Diary

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Press, Study Director — Neuren Pharmaceuticals
Locations (4):
- United States (4):
  - Rady Children's Hospital San Diego, San Diego, California
  - Rare Disease Research, Atlanta, Georgia
  - Uncommon Cures, Chevy Chase, Maryland
  - Suburban Research, Media, Pennsylvania

IPD SHARING:
Plan to Share IPD: No